CLINICAL TRIAL: NCT02890368
Title: A Phase 1 Dose Escalation Trial of Intratumoral Injections of TTI-621 in Subjects With Relapsed and Refractory Percutaneously-Accessible Solid Tumors and Mycosis Fungoides
Brief Title: Trial of Intratumoral Injections of TTI-621 in Subjects With Relapsed and Refractory Solid Tumors and Mycosis Fungoides
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTI-621-02
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumors; Mycosis Fungoides; Melanoma; Merkel-cell Carcinoma; Squamous Cell Carcinoma; Breast Carcinoma; Human Papillomavirus-Related Malignant Neoplasm; Soft Tissue Sarcoma
Keywords: CD47; SIRPa; Immunotherapy; Checkpoint inhibitor
MeSH Terms: conditions — Mycosis Fungoides; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Squamous Cell; Breast Neoplasms; Sarcoma | interventions — TTI-621; talimogene laherparepvec; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- TTI-621 Monotherapy Escalation (Experimental): TTI-621 Escalation phase of single or multiple doses of TTI-621 delivered by intratumoral injections (various dose cohorts).
  Interventions: Drug: TTI-621 Monotherapy
- TTI-621 Monotherapy (Single Lesion) (Experimental): TTI-621 Single Lesion Injection Expansion Cohort
  Interventions: Drug: TTI-621 Monotherapy
- TTI-621 Monotherapy (Multiple Lesions) (Experimental): TTI-621 Multiple Lesion Injections Expansion Cohort
  Interventions: Drug: TTI-621 Monotherapy
- TTI-621 + PD-1/PD-L1 Inhibitor (Experimental): Combination Therapy Expansion Cohort of TTI-621 plus PD-1/PD-L1 Inhibitor
  Interventions: Drug: TTI-621 + PD-1/PD-L1 Inhibitor
- TTI-621 + Pegylated Interferon-α2a (Experimental): Combination Therapy Expansion Cohort of TTI-621 plus Pegylated Interferon-α2a
  Interventions: Drug: TTI-621 + pegylated interferon-α2a
- TTI-621 + T-Vec (Experimental): Combination Therapy Expansion Cohort of TTI-621 plus T-Vec
  Interventions: Other: TTI-621 + T-Vec
- TTI-621 + Radiation (Experimental): Combination Therapy Expansion Cohort of TTI-621 plus Radiation Therapy
  Interventions: Other: TTI-621 + radiation

INTERVENTIONS:
Drug: TTI-621 Monotherapy — TTI-621 (SIRPα-IgG1 Fc) is a soluble recombinant fusion protein created by directly linking the sequences encoding the N-terminal CD47 binding domain of human SIRPα with the Fc domain of human immunoglobulin (IgG1). TTI-621 acts by binding human CD47 and preventing it from delivering an inhibitory "do not eat" (antiphagocytic) signal to macrophages.
  Other Names: SIRPα-IgG1 Fc
  Arms: TTI-621 Monotherapy (Multiple Lesions); TTI-621 Monotherapy (Single Lesion); TTI-621 Monotherapy Escalation
Drug: TTI-621 + PD-1/PD-L1 Inhibitor — TTI-621 will be given in combination with one of the following programmed death-1 (PD-1) or programmed death-ligand-1 (PD-L1) inhibitors: nivolumab, pembrolizumab, durvalumab, avelumab, or atezolizumab administered on Day 1. Subjects in this cohort must have a cancer diagnosis for which a PD-1/PD-L1 inhibitor is approved by the FDA or listed in the National Comprehensive Cancer Network (NCCN) Guidelines.
  Other Names: SIRPα-IgG1 Fc + PD-1/PD-L1 Inhibitor
  Arms: TTI-621 + PD-1/PD-L1 Inhibitor
Drug: TTI-621 + pegylated interferon-α2a — TTI-621 will be given in combination with pegylated interferon-α2a. Subjects in this cohort must have a cancer diagnosis for which pegylated interferon-α2a is approved by the FDA or listed in the National Comprehensive Cancer Network (NCCN) Guidelines.
  Other Names: SIRPα-IgG1 Fc + pegylated interferon-α2a
  Arms: TTI-621 + Pegylated Interferon-α2a
Other: TTI-621 + T-Vec — TTI-621 will be given in combination with talimogene laherparepvec (T-Vec). Subjects in this cohort must have unresectable melanoma.
  Other Names: SIRPα-IgG1 Fc + talimogene laherparepvec
  Arms: TTI-621 + T-Vec
Other: TTI-621 + radiation — TTI-621 will be given following radiation to the target plasmacytoma. Subjects in this cohort must have relapsed multiple myeloma with bony or soft tissue plasmacytoma(s).
  Other Names: SIRPα-IgG1 Fc + radiation
  Arms: TTI-621 + Radiation

SUMMARY:
This is a multicenter, open-label, phase 1 study conducted to test intratumoral injections of TTI-621 in subjects that have relapsed and refractory percutaneously accessible solid tumors or mycosis fungoides.

The study will be performed in two different parts. Part 1 is the Dose Escalation phase and Part 2 is the Dose Expansion phase.

The purpose of this study is to characterize the safety profile of TTI-621 and to determine the optimal dose and delivery schedule of TTI-621. In addition, the safety and antitumor activity of TTI-621 will be evaluated in combination with other anti-cancer agents or radiation.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase 1 study conducted to test intratumoral injections of TTI-621 in patients that have relapsed and refractory percutaneously accessible solid tumors or mycosis fungoides.

TTI-621 (SIRPα-IgG1 Fc) is a soluble recombinant fusion protein created by directly linking the sequences encoding the N-terminal CD47 binding domain of human SIRPα with the Fc domain of human immunoglobulin (IgG1). TTI-621 acts by binding human CD47 and preventing it from delivering an inhibitory "do not eat" (antiphagocytic) signal to macrophages.

The study will be performed in two different parts: Dose Escalation and Dose Expansion.

During the escalation part of the study, TTI-621 was studied at 3 different dose levels and at different dosing frequencies to characterize safety, tolerability, pharmacokinetics, and to determine the maximum tolerated dose (MTD).

During the expansion part of the study, TTI-621 will be studied in an expanded group of patients at the maximum feasible dosing regimen determined in the escalation phase. After completion of their initial assigned therapy, subjects may receive continuation with TTI-621. The expansion phase will further define safety and characterize efficacy of TTI-621 alone and in combination with other anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, injectable cancer lesion (limited to solid tumors and mycosis fungoides)
* Adequate renal function
* Adequate coagulation function
* Adequate hepatic function
* Disease that has progressed on standard therapy or for whom there is no other therapy option available

Exclusion Criteria:

* Central nervous system involvement
* Significant cardiovascular disease
* Active autoimmune disease
* Active hepatitis B or C or a history of HIV infection
* Uncontrolled infection
* History of hemolytic anemia or bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Optimal TTI-621 delivery regimen | 10 months
  Defining the optimal TTI-621 delivery regimen in subjects with advanced percutaneously-accessible cancer

SECONDARY OUTCOMES:
Frequency and severity of adverse events | 15 months
  Safety of TTI-621 when given to subjects with relapsed and refractory percutaneously-accessible solid tumors and Mycosis Fungoides alone and in combination with other anti-cancer drugs or radiation
Preliminary evidence of anti-tumor activity of TTI-621 | 15 months
  Preliminary evidence of anti-tumor activity of TTI-621 when given to subjects with relapsed and refractory percutaneously-accessible solid tumors and Mycosis Fungoides alone and in combination with other anti-cancer drugs or radiation

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Querfeld C, Thompson JA, Taylor MH, DeSimone JA, Zain JM, Shustov AR, Johns C, McCann S, Lin GHY, Petrova PS, Uger RA, Molloy N, Shou Y, Akilov OE. Intralesional TTI-621, a novel biologic targeting the innate immune checkpoint CD47, in patients with relapsed or refractory mycosis fungoides or Sezary syndrome: a multicentre, phase 1 study. Lancet Haematol. 2021 Nov;8(11):e808-e817. doi: 10.1016/S2352-3026(21)00271-4. Epub 2021 Oct 7. PMID 34627593
- [Derived] Kruglov O, Johnson LDS, Minic A, Jordan K, Uger RA, Wong M, Sievers EL, Shou Y, Akilov OE. The pivotal role of cytotoxic NK cells in mediating the therapeutic effect of anti-CD47 therapy in mycosis fungoides. Cancer Immunol Immunother. 2022 Apr;71(4):919-932. doi: 10.1007/s00262-021-03051-x. Epub 2021 Sep 14. PMID 34519839